CLINICAL TRIAL: NCT02749422
Title: A Randomized Controlled Pilot Study of TMS Enhancement of Associative Memory Networks in Healthy Subjects and Epilepsy Patients
Brief Title: fMRI Guided TMS Enhancement of Associative Memory Networks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was closed prematurely due to longer-than-expected recruitment times.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-00732
Record Dates: First submitted 2016-04-13; First posted 2016-04-25 (Estimated); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy
Keywords: cognitive dysfunction; memory loss; non-invasive transcranial magnetic stimulation (TMS); rTMS; Magstim Rapid2
MeSH Terms: conditions — Epilepsy; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Healthy Subjects (Active Comparator)
  Interventions: Diagnostic Test: MagStim RapidStim2
- Temporal Lobe Epilepsy Patients (Experimental)
  Interventions: Diagnostic Test: MagStim RapidStim2

INTERVENTIONS:
Diagnostic Test: MagStim RapidStim2 — Repetitive transcranial magnetic stimulation (TMS)

SUMMARY:
This is a randomized, single-blinded, controlled phase 1 study to demonstrate feasibility and explore the neurophysiologic and clinical effects of repetitive transcranial magnetic stimulation (TMS) interventions in epilepsy patients and healthy controls. The inclusion of a control group will be used to see whether epilepsy patients, who suffer from a higher degree of comorbid memory difficulty presumably from entorhinal-hippocampal dysfunction, can benefit from a TMS intervention can benefit as much as a healthy matched population. Investigators will also be looking at functional connectivity between the hippocampus and cortical regions

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Right-handed
* Score at least 26 out of 30 on the Montreal Cognitive Assessment (MOCA). Healthy subjects will be matched to age, handedness, and education compared to epilepsy subjects.
* Must be able to provide informed consent.

Exclusion Criteria:

* Any history of a neurological disorder
* Chronic or progressive medical condition
* Any history of severe traumatic brain injury or skull defect
* Metal or devices in the head, including neurostimulators of metal foreign bodies
* Any other implanted metal device, including pacemaker, spinal cord stimulator, VNS.
* Any other ferromagnetic substance in the body (including tattoos, dental prosthetics, etc).
* Taking a medication which may lower the seizure threshold within the 4 weeks prior to the start of the study, including use of neuroleptic (esp. clozapine), antibiotic (penicillin, cephalosporins), and bronchodilating medications.
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anli Liu, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patients were enrolled in the Healthy Subjects arm.
Period: Overall Study
Arm/Group | Healthy Subjects | Temporal Lobe Epilepsy Patients
Started | 0 | 8
Completed | 0 | 5
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled in the "Healthy Subject" study arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Subjects | Temporal Lobe Epilepsy Patients | Total
Number analyzed (Participants) | 0 | 5 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 26.6 (7.3) | 26.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 4 | 4
  Male |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 1 | 1
  Unknown or Not Reported |  | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Face-Object Pair Association Task Score During Left Lateral Parietal Site Stimulation
Description: A face-object pair association task will be administered before and after rTMS treatment at each treatment session. This measure is evaluating the mean change in the task score from immediately before rTMS is applied to the left lateral parietal site to immediately after treatment.
Time Frame: Immediately before Left Lateral Parietal Site Stimulation, Immediately after Left Lateral Parietal Site Stimulation (20 minute procedure; Up to Week 6)
Population: Data for this outcome measure were not collected from participants in the study.
Arm/Group | Healthy Subjects | Temporal Lobe Epilepsy Patients
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Mean Change in Face-Object Pair Association Task Score During Motor Cortex Stimulation
Description: A face-object pair association task will be administered before and after rTMS treatment at each treatment session. This measure is evaluating the mean change in the task score from immediately before rTMS is applied to the motor cortex to immediately after treatment.
Time Frame: Immediately before Motor Cortex Stimulation, Immediately after Motor Cortex Stimulation (20 minute procedure; Up to Week 6)
Population: Data for this outcome measure were not collected from participants in the study.
Arm/Group | Healthy Subjects | Temporal Lobe Epilepsy Patients
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in fMRI-based Functional Connectivity Between Hippocampus and Cortical Regions
Description: Changes in hippocampal-cortical functional connectivity will be identified using voxel-wise paired T-tests. The change will be measured between baseline assessment and resting state fMRI assessment following rTMS.
Time Frame: Baseline, Week 6
Population: Data for this outcome measure were not collected from participants in the study.
Arm/Group | Healthy Subjects | Temporal Lobe Epilepsy Patients
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Change in Word-Pair Association Task Score During Left Lateral Parietal Site Stimulation
Description: A word-pair association task will be administered before and after rTMS treatment at each treatment session. This measure is evaluating the mean change in the task score from immediately before rTMS is applied to the left lateral parietal site to immediately after treatment.
Time Frame: as for outcome 1
Population: Data for this outcome measure were not collected from participants in the study.
Arm/Group | Healthy Subjects | Temporal Lobe Epilepsy Patients
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Change in Word-Pair Association Task Score During Motor Cortex Stimulation
Description: A word-pair association task will be administered before and after rTMS treatment at each treatment session. This measure is evaluating the mean change in the task score from immediately before rTMS is applied to the motor cortex to immediately after treatment.
Time Frame: as for outcome 2
Population: Data for this outcome measure were not collected from participants in the study.
Arm/Group | Healthy Subjects | Temporal Lobe Epilepsy Patients
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 months
Description: No subjects were enrolled in the "Healthy Subjects" arm; the number of participants at risk is zero for this arm.
Arm/Group | Healthy Subjects | Temporal Lobe Epilepsy Patients
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/5
Other Adverse Events (participants affected / at risk) | 0/0 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT02749422/Prot_SAP_000.pdf